CLINICAL TRIAL: NCT03100201
Title: Robotic-assisted Training After Upper Arm Fracture - a Multicentre, Controlled and Randomized Intervention Study
Brief Title: Robotic-assisted Training After Upper Arm Fracture
Acronym: RASTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Collaborators: BG Unfallklinik Murnau (Other); Berufsgenossenschaftliche Unfallklinik Ludwigshafen (Other); Deutsche Gesetzliche Unfallversicherung (DGUV) (Unknown)
Responsible Party: Principal Investigator, Corinna Nerz, Research associate, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RASTA 2016
Record Dates: First submitted 2017-03-22; First posted 2017-04-04 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Shoulder Injury
Keywords: robotic-assisted rehabilitation; humeral fracture; randomised controlled study
MeSH Terms: conditions — Shoulder Injuries; Humeral Fractures | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Patients will be recruited in three different clinics in Germany and randomised into an intervention and a control group. All patients will receive conventional occupational- and physiotherapy. The intervention group will receive an additive robotic-assisted training using the Armeo®Spring robot for three weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Armeo®Spring (Active Comparator): The intervention group will receive conventional occupational- and physiotherapy and an additive robotic-assisted training using the Armeo®Spring robot for three weeks.
  Interventions: Other: Intervention Armeo®Spring
- Control group (Active Comparator): The control group will receive conventional occupational- and physiotherapy.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Intervention Armeo®Spring — The robotic-assisted training will be performed using the clinically evaluated Armeo®Spring medical device (Hocoma AG, Zurich, Switzerland). By means of a sensory orthosis, arm movements will be supported and transmitted to a computer system and visually shown on a screen.
  Arms: Intervention Armeo®Spring
Other: Control Group — The control group will receive conventional occupational- and physiotherapy over 3 weeks
  Arms: Control group

SUMMARY:
In this study, patients with upper arm fracture will receive an additive robotic-assisted training using the Armeo®Spring robot for three weeks on the injured arm in addition to conventional physio- and occupational therapy. The supportive treatment and execution of specific exercises on the Armeo®Spring should lead to improved recovery of function and mobility of the upper arm compared to conservatively treated patients.

DETAILED DESCRIPTION:
60 Patients aged between 35 and 70 years with proximal humeral fracture and surgical treatment will be recruited in three different clinics in Germany and randomised into an intervention and a control group. Participants will be assessed before randomisation and followed up after completing an intervention period of 3 weeks and additionally after 3, 6 and 12 months. Baseline assessment will assess cognition (SOMC), level of pain in the affected arm, ability to work, gait speed (10m walk), disability of the arm, shoulder and hand (DASH), as well as the range of motion of the affected arm (goniometer measurement), visual acuity and motor function of orthopaedic patients (WMFT-O). Clinical follow up directly after intervention will assess disability of the arm, shoulder and hand (DASH), the range of motion and motor function (WMFT-O). Primary outcome parameter will be the DASH and secondary outcome parameter will be the WMFT-O. The long-term results will be assessed prospectively by a postal follow-up. All patients will receive conventional occupational- and physiotherapy. The intervention group will receive an additive robotic-assisted training using the Armeo®Spring robot for three weeks.

ELIGIBILITY:
Inclusion Criteria:

* surgical treatment of the shoulder joint after upper arm fracture classified as type AO 11
* movement-stable fracture
* Inclusion between the fourth and the seventh week after surgery

Exclusion Criteria:

* limited cognition as defined by a score in Short-Orientation-Memory-Concentration Test (SOMC) less than 10 points
* inadequate level of pain during movement of the affected shoulder joint (pain score >5 on a visual analogue pain scale)
* strongly limited vision or hearing
* heart failure (New York Heart Association stage III-IV) or COPD (Chronic Obstructive Pulmonary Disease) Gold stage III-IV
* walking speed <0.8m/sec
* isolated tuberculum majus fracture of the humerus (AO 11, A1)
* fractures with involvement of the glenoid cavity
* double fractures
* injury of the plexus or the axillaris nerve

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in disability of the arm, shoulder and hand (DASH) | DASH will be assessed before randomisation and followed up after completing an intervention period of 3 weeks and additionally after 3, 6 and 12 months for assessing the change
  subjective questionnaire for assessing the disability of the arm, shoulder and hand

SECONDARY OUTCOMES:
Change in the WMFT-O | WMFT will be assessed before randomisation and followed up after completing an intervention period of 3 weeks for assessing the change
  WMFT-O is an objective test for assessing the disability of the shoulder
Change in ROM | ROM will be assessed before randomisation and followed up after completing an intervention period of 3 weeks for assessing the change
  a goniometer-based measurement of the active range of motion (ROM) of the shoulder joint
Change in grip strength | grip strength will be assessed before randomisation and followed up after completing an intervention period of 3 weeks for assessing the change
  measurement of the grip strength using the Jamar dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Peter Augat, Prof., Study Chair — BG Unfallklinik Murnau
Locations (3):
- Germany (3):
  - Berufsgenossenschaftliche Klinik Ludwigshafen, Ludwigshafen
  - Berufsgenossenschaftliche Klinik Murnau, Murnau am Staffelsee
  - Robert-Bosch-Hospital, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022 Jun 21;6(6):CD000434. doi: 10.1002/14651858.CD000434.pub5. PMID 35727196
- [Derived] Nerz C, Schwickert L, Scholch S, Gordt K, Nolte PC, Kroger I, Augat P, Becker C. Inter-rater reliability, sensitivity to change and responsiveness of the orthopaedic Wolf-Motor-Function-Test as functional capacity measure before and after rehabilitation in patients with proximal humeral fractures. BMC Musculoskelet Disord. 2019 Jul 6;20(1):315. doi: 10.1186/s12891-019-2691-0. PMID 31279331
- [Derived] Nerz C, Schwickert L, Becker C, Studier-Fischer S, Mussig JA, Augat P. Effectiveness of robot-assisted training added to conventional rehabilitation in patients with humeral fracture early after surgical treatment: protocol of a randomised, controlled, multicentre trial. Trials. 2017 Dec 6;18(1):589. doi: 10.1186/s13063-017-2274-z. PMID 29212528